CLINICAL TRIAL: NCT01754038
Title: Patients Receiving Integrative Medicine Interventions Effectiveness Registry
Brief Title: Registry for Integrative Medicine Interventions Effectiveness
Acronym: PRIMIER
Status: Completed | Type: Observational
Sponsor: BraveNet (Other)
Collaborators: The Bravewell Collaborative (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00040886
Record Dates: First submitted 2012-12-17; First posted 2012-12-21 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: All Conditions of Integrative Medicine Clinic Patients
Keywords: Patient Reported Outcomes; PRO; Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Integrative Medicine Clinic Attendees: All patients attending a participating Integrative Medicine clinic for clinical services will be invited to participate in the PRIMIER Registry

SUMMARY:
This registry will perform prospective surveillance of participants attending collaborating Integrative Medicine clinic sites for clinical services. All decisions about medication use, treatments, visit frequency, assessment of tolerance, and other aspects of patient management will be left to the clinical providers' discretion. We will attempt to follow the participants in the PRIMIER Registry for up to 2 years.

Essential data elements that capture patient-reported outcomes and measures of clinical activity will be obtained at approximately 2-month intervals for the first 6 months, then every 6 months through the end of year 2.

DETAILED DESCRIPTION:
Rationale:

According to the Agency for Healthcare Research and Quality (AHRQ), observational databases provide an opportunity for simultaneous exploration of the impact of integrative medicine on various medical conditions. As opposed to selecting a single condition for which patients may seek care at our sites, the project will allow us to collect prospective patient-reported outcomes on a number of frequently seen medical conditions. By clustering participants at the multiple IM clinical sites with the same medical condition, we will be able to compare the impact of various integrative therapies on patient-reported outcomes.

Objectives:

Primary Objective

1. To evaluate the change in patient-reported outcomes (e.g. quality of life, mood and stress) over time

Secondary Objectives

1. To evaluate whether patient-reported outcomes differ by baseline characteristics of the participants (e.g. demographics, clinical condition, intervention sought)
2. In a subset of clinics, to collect cost data from patient encounters to allow cost comparisons among the interventions and outcomes

OUTCOME ASSESSMENTS Patient Reported Outcomes (PROs) The PRIMIER Registry will use the Research Electronic Data Capture (REDCap) as an online research management tool that can be used to collect PRO data. REDCap is a free, online research management tool that enables researchers to create study-specific Web sites for capturing participant data securely.

Patient-Reported Outcomes (PROs) is the term used to denote health data that is provided by the patient through a system of reporting. A PRO is basically a patient's feedback on their feelings or functions as they are dealing with chronic diseases or conditions. PROs can also be measured when patients are undergoing treatment or are participating in a clinical trial.

The Patient-Reported Outcome Measurement Information System (PROMIS®), funded by the National Institutes of Health, aims to provide clinicians and researchers access to efficient, valid, and responsive self-reported measures of health, including symptoms, function and well-being. PROMIS® instruments (short forms, computerized adaptive tests (CATs), profiles) are a central feature of the Assessment Center instrument library.

PROMIS® is unique from other PRO systems in four ways:

1. PROMIS® data is comparable because there are common measurements across domains
2. PROMIS® measures are reliable and valid. They have been subjected to rounds of rigorous review and testing to ensure that the measurements are precise, consistent, and accurate.
3. PROMIS® is flexible: PRO tools or measures can be obtained by way of in-person interviews, written questionnaires or computer-assisted tools.
4. PROMIS® is inclusive in that all people regardless of literacy, language, physical function and life status can use its tools

The PRIMIER Registry will use the PROMIS-29 as the core data PRO collection tool along with the Perceived Stress Scale-4 (PSS-4)and the Patient Activation Measure (PAM).

Cost Indicators

In a subset of sites, we will collect cost indicators of healthcare resource utilization, including prescription medications, over-the-counter medications, physician and ER visits, as well as measures of patient functionality such as work productivity. This analysis will use the treatment utilization data obtained from the patient visit questionnaires as these data allowed us to count the specific number of treatments each patient reported over the course of the study. Patients will be asked to report the number of each type of IM treatment session received at every data collection time point. In the event that a patient skipped an interim study visit, they will be asked to report cumulative counts of IM treatment sessions received since their previous visit. We recognize that patients may not readily recall this information, so to ensure accuracy of this measure, research coordinators (or other research staff) will review the patients' medical record to quantify the type and number of visits to the participating integrative medicine clinical sites during study participation.

Statistical Design

Primary Analysis The main analyses of the PRIMIER Registry will be descriptive and summary.

Major Secondary Analyses Since the PRIMIER Registry will collect many of the same variables over a 2 year period, the secondary analyses will include examining the repeated variables and changes from baseline.

General Statistical Methods We will summarize descriptive statistics using frequencies (percentages) for categorical variables. We will report means, standard deviations, medians, quartiles, minimums, and maximums for all continuous variables.

We will use univariate analyses to detect outliers which will be subsequently submitted as queries to sites to ensure clean data. Questionnaires that can be aggregated into a score will be scored and the scores will be used for summarizing.

We will perform repeated-measures analyses of variance to detect changes in PRO and cost indicators over time. We will summarize results with a point estimate of mean change in the outcome measures between baseline and any specified follow-up visit with 95% confidence intervals. We will report P values for overall model summary, indicating any difference between any two given points. If the P value is significant (<0.05), we will perform follow-up linear regression analyses to verify that the trends are consistent in direction throughout all study visits, indicating constant improvement or decline from visit to visit.

Exploratory Analyses We will look for variables and trends that are of interest to the collaborating investigators to explore. The appropriate analysis plan will be developed to take advantage of the wealth of data that will be collected in the PRIMIER Registry. At this time, we do not know what future analyses will be conducted.

We do not know the medical conditions for which individual participants in this PRIMIER Registry will seek help at the IM clinic, nor will we know in advance which IM interventions patients will receive. With these limitations, we cannot predefine subgroups for statistical analyses at present. However, in the future we will define post-hoc groups by clinical condition (e.g., participants with cancer, chronic pain, headaches, etc.) or IM intervention received (e.g., acupuncture, meditation, massage, etc.) for further analyses.

ELIGIBILITY:
Inclusion Criteria:

* Be seen as a clinical patient in one of the participating Integrative Medicine (IM) clinics and willing to participate in the Registry
* Be 18 years of age or older
* Have access to a computer with internet connection and a valid email address
* Be willing to be contacted in the future by study investigators

Exclusion Criteria:

* Not being seen by a provider for clinical purposes, but only involved in an education program or one-time activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients attending a participating Integrative Medicine Clinic
Sampling Method: Non-Probability Sample
Enrollment: 5069 (Actual)
Dates: Start 2013-08; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
PROMIS® CAT | Baseline, 2, 4, 6 months, then every 6 months through year 2,.
  PROMIS® can integrate Item Response Theory (IRT) with computers to administer a PRO instrument. IRT selects questions on the basis of a patient's response to previously administered questions, measurement is "adapted" to individual, skips uninformative items to minimize response burden and allows determination of person's standing on a domain without a loss in measurement precision. The PROMIS® CAT for PRIMIER will be designed to assess anxiety, depression, sleep disturbance, fatigue, pain interference, physical function, and satisfaction with participation in social roles. Questions will be answered electronically using a standard 1-5 Likert scale. Participants will answer between 4 and 12 questions per domain, for a total of 29 to 85 questions.

SECONDARY OUTCOMES:
Perceived Stress Scale - 4 | Baseline, 2, 4, 6 months, then every 6 months through year 2.
  The PSS-4 is brief, validated and widely used psychological instrument for assessing a participant's perception of stress change. The PSS-4 consists of 4 questions to measure the degree to which situations in the participant's life are perceived as stressful including questions related to perceived unpredictability and lack of control. Participants choose responses ranging from never (0) to very often (4) with a total score ranging from 0 to 16.
Patient Activation Measure (PAM) | Baseline, 2, 4, 6 months, then every 6 months through year 2.
  The PAM is a brief, validated instrument for gauging the knowledge, skills and confidence essential to managing one's own health and healthcare. The 13-item PAM assessment segments consumers into one of four progressively higher activation levels. Each level addresses a broad array of self-care behaviors and offers deep insight into the characteristics that drive health activation.
Cost Indicators | Every 6 months
  From the subjects' medical and financial records we will capture ICD codes, CPT codes, and payments made by subjects and their insurance companies.

CONTACTS AND LOCATIONS:
Overall Officials: Donald I Abrams, MD, Principal Investigator — University of California, San Francisco; Jeffrey A Dusek, PhD, Principal Investigator — Penny George Institute for Health and Healing, Abbott Northwestern Hospital; Diane McKee, MD MS, Study Director — Albert Einstein College of Medicine
Locations (14):
- United States (14):
  - Scripps Center for Integrative Medicine, La Jolla, California
  - UCSF Osher Center for Integrative Medicine, San Francisco, California
  - Venice Family Clinic at Simms/Mann Health and Wellness Center, Santa Monica, California
  - University of Colorado School of Medicine, Center for Integrative Medicine, Aurora, Colorado
  - Northwestern Integrative Medicine - Northwestern Memorial Physicians Group, Chicago, Illinois
  - University of Maryland Center for Integrative Medicine, Baltimore, Maryland
  - Program for Integrative Medicine and Health Care Disparities, Boston, Massachusetts
  - Penny George Institute for Health and Healing, Minneapolis, Minnesota
  - Beth Israel Integrative Medicine Continuum Center for Health and Healing, New York, New York
  - Duke Integrative Medicine Clinic, Durham, North Carolina
  - Alliance Institute for Health and Healing, Cincinnati, Ohio
  - Jefferson-Myrna Brind Center of Integrative Medicine, Philadelphia, Pennsylvania
  - UPMC Shadyside Center for Integrative Medicine, Pittsburgh, Pennsylvania
  - Vanderbilt Center for Integrative Health, Nashville, Tennessee

REFERENCES:
- [Derived] Dusek JA, Gao Q, Kim RS, Abrams DI, Kligler B, Dyer NL, Hansen K, Roseen EJ, McKee MD; PRIMIER Writing Group*. Patients Receiving Integrative Medicine Effectiveness Registry (PRIMIER) of the BraveNet practice-based research network: Results of the chronic pain cohort. Integr Med Res. 2025 Jun;14(2):101141. doi: 10.1016/j.imr.2025.101141. Epub 2025 Mar 25. PMID 40297756
- [Derived] Dusek JA, Abrams DI, Roberts R, Griffin KH, Trebesch D, Dolor RJ, Wolever RQ, McKee MD, Kligler B. Patients Receiving Integrative Medicine Effectiveness Registry (PRIMIER) of the BraveNet practice-based research network: study protocol. BMC Complement Altern Med. 2016 Feb 4;16:53. doi: 10.1186/s12906-016-1025-0. PMID 26846166